CLINICAL TRIAL: NCT04079244
Title: Analysis of the Link Between Flow State and Preoperative Anxiety in Children Undergoing Playful Distraction - Studying the Benefits of Digital Distractions in an Ambulatory Care Service
Brief Title: Analysis of the Link Between Flow State and Preoperative Anxiety in Children Undergoing Playful Distraction
Acronym: ALFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: University of Rennes 2 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC19_30028_ALFA
Record Dates: First submitted 2019-08-30; First posted 2019-09-06 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Children; Ambulatory Surgery; General Anesthesia
Keywords: Preoperative anxiety; Distractions; Flow; Child

STUDY DESIGN:
Intervention Model Description: The attribution to the game-video or cartoon group is carried out according to a randomization by block " week ".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video game (Active Comparator): Children receive a tablet with a video game at their arrival on the unit until the introduction of the anesthesia mask.
  The video game used is "Le Héros C'est Toi", a game specially developed for the unit. The game recreates the hospital environment and includes mini-games geared to children
  Interventions: Behavioral: Video game
- Animated cartoon (Active Comparator): Children receive a tablet with an animated cartoon at their arrival on the unit until the introduction of the anesthesia mask.
  The cartoon used is "L'âge de glace", an animated cartoon geared to children.
  Interventions: Behavioral: Animated cartoon

INTERVENTIONS:
Behavioral: Video game — Children receive a tablet with a video game at their arrival on the unit until the introduction of the anesthesia mask.
  The video game used is "Le Héros C'est Toi", a game specially developed for the unit. The game recreates the hospital environment and includes mini-games geared to children.
  Arms: Video game
Behavioral: Animated cartoon — Children receive a tablet with an animated cartoon at their arrival on the unit until the introduction of the anesthesia mask.
  The cartoon used is "L'âge de glace", an animated cartoon geared to children.
  Arms: Animated cartoon

SUMMARY:
This study focuses on preoperative anxiety in children and non-drug methods to reduce anxiety.

During surgery under general anesthesia, children may be anxious because of separation from their parents, fear of anesthesia, or loss of control.

In order to reduce the anxiety of the child, anesthesiologists sometimes use an anxiolytic medicine. This premedication can reduce the anxiety of children. However, side effects are often observed as rebound anxiety after the operation or a delay to discharge from hospital.

In recent years, alternative methods to premedication have been studied to reduce the anxiety of children. For example, video games and cartoons are distraction methods. Studies have shown that using a video game or cartoon during the waiting phases (in the room, when traveling, in the permutation room) reduces the anxiety of children and with the same efficiency as anxiolytic.

In this study, the investigators will evaluate the effectiveness of a tablet game and a cartoon to reduce the anxiety of children.

DETAILED DESCRIPTION:
This study takes an interest on the problem of the well-being of children during an outpatient surgery.

Children are often anxious before a surgery under general anesthetic because of unfamiliar environments, separation from parents, loss of control or uncertainty about anesthesia. 50% to 70% of children develop anxiety after surgery. Anxiety before surgery are associated with behavioral changes in postoperative like increase in anxiety, sleep or eating disturbances and with postoperative pain.

To reduce this preoperative anxiety, the use of anxiolytics (hypnovel, hydroxizyne) is the most commonly used method. But this premedication remains controversial (paradoxical effects with rebound of anxiety, loss of explicit memorization).

The aim of this study is to examine two non-pharmacological and non-invasive methods (technological distraction through video games and animated cartoons) that seem to be effective in reducing preoperative anxiety and its postoperative repercussions. Much studies show the benefits of preoperative distraction method to reduce children's anxiety, such as cartoons, video games, puzzles.

It is now necessary to understand the processes underlying the relationship between the preoperative anxiety and distraction method.

Video games and cartoons are supposed to foster a high level of cognitive engagement in children, which would allow them to focus less on the anxiogenic elements of the operating context and thus reduce their preoperative anxiety. This state of cognitive engagement is called flow. Flow is defined as a state in which person is so involved in an activity that nothing else matters.

Within the paediatric anaesthesia department of the University Hospital Rennes Sud, the playful video game "Le Héros C'est Toi" is systematically offered to children aged 3 to 10 years to accompany them throughout the course of care during outpatient surgery. This has been a standard practice since 2014.

In this project, the aim is to examine the links between the state of flow, generated by a playful application on tablet or animated cartoon, and the preoperative anxiety of children.

Protocol :

The day of the intervention surgery, the study is proposed to the parents and the children on their arrival. If the participants are in favor, the consent documents are given to them. Patient inclusion is ongoing, after verification of inclusion criteria, parental consent and signed consent. The attribution to the game-video or cartoon group is carried out according to a randomization by block " week ".

At their arrival in ambulatory care service, when child is in the room a first video recording is made in order to examine the anxiety of the child. Then tablet with the video game or animated cartoon is made available to the child. The tablet is available to the child until anesthetic induction.

Four others video recording are made :

* before the child leaves for the waiting room to examine the flow state of the child until the separation with the parents to examine the anxiety of the child,
* when the child is in the waiting room to examine the flow state of the child
* and during the anesthetic induction to examine the anxiety of the child.

While the children are in the operating room, parents must complete questionnaires to evaluate anxiety-trait of the children and anxiety-state of the parent.

The pain's score and the emergence delirium of the child on waking are recorded.

The day after the intervention, a call is made to parents to examine the postoperative behavioral changes of the children. Two other calls are made a week after and a month after.

Materials:

To examine the anxiety-state of the child on video recording the investigators use an observational grid, the mYPAS To examine the anxiety-trait of the child the investigators use the questionnaire PAS-R To examine the anxiety-state of the parents the investigators use the questionnaire STAI-S To examine the pain of the child on waking the investigatorsuse an observational grid FLACC To examine the emergence delirium of the child on waking the investigators use an observational grid, the EPAD To examine the flow state on video recording of the child, the investigatorsuse an observational grid. This tool is currently psychometrically tested.

To examine the postoperative behavioral change, the investigators use the questionnaire PHBQ

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 10 years
* Benefiting from an ambulatory surgery under general anesthesia
* Whose parents or the legal representative of the parental authority do not object to his participation
* Written consent of one of the parents or the legal representative of the parental authority to the video recording of the child.

Exclusion Criteria:

* Children participating in another study
* No understanding of the French language by the parents and/or the child
* Major developmental delay, psychiatric pathology or visual impairment that does not allow the children to play on a tablet.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2019-09-28 (Actual)

PRIMARY OUTCOMES:
correlation between the flow state and preoperative anxiety | On the day of surgery
  This will involve assessing the correlation between the flow state and preoperative anxiety.
  The tool used is the mYPAS. It is an observation based-method. Observation grid is composed of five dimensions : activity, vocalizations, emotional expressivity, state of apparent arousal, use of parents. The observer chooses a score for the five dimensions based on the criteria provided in the grid.
  The tool used is the Flow Observation Grid. It is an observation based-method. Observation gri dis composed of three dimensions : concentration, joy, frustration. The observer chooses a score for the three dimensions based on the criteria provided in the grid.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wodey, PH-PD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France